CLINICAL TRIAL: NCT07143305
Title: Effect of Citrulline Malate Supplementation During a Multicomponent Exercise Program on Physical Function and Biochemical Parameters in Physically Active Older Women: a Randomised Controlled Pilot Trial
Brief Title: Effect of Citrulline Malate Supplementation on Physical Function and Biochemical Parameters in Physically Active Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Principal Investigator, Juan Francisco Mielgo, Principal Investigator, Universidad de Burgos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CITMAL
Record Dates: First submitted 2025-08-08; First posted 2025-08-27 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-08

CONDITIONS: Supplementation
Keywords: citrulline; Physical Performance; older women

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Active Comparator): Placebo supplementation with 3 g/day of maltodextrine
  Interventions: Other: Multicomponent physical exercise programme
- Supplementation (Experimental): 3 g/day of citrulline malate
  Interventions: Other: Multicomponent physical exercise programme

INTERVENTIONS:
Other: Multicomponent physical exercise programme — Participants engaged in a multicomponent physical exercise programme designed specifically for older adults. The programme was based on the latest evidence and international recommendations for sarcopenia and functional maintenance in ageing population.

SUMMARY:
A randomised, double-blind, placebo-controlled pilot trial was conducted with thirty-three community-dwelling women aged 65 years or over. Participants were assigned to a multicomponent training programme (three days per week) and received either 3 g per day of citrulline malate or a placebo. Assessments were conducted before and after the intervention, including tests of physical performance (6MWT, sit-to-stand, SPPB), blood biomarkers (vitamin D, glucose, CK, hormones), and perceived quality of life (WHOQOL-BREF).

ELIGIBILITY:
Each participant underwent a comprehensive medical evaluation by their primary care physician to confirm their health status and eligibility.

Inclusion criteria:

* Sex: women.
* Age: 60-75 years.

Exclusion criteria:

* Functional limitations (Barthel Index <100 and/or Lawton-Brody Scale <8).
* Musculoskeletal injuries within the past six months.
* Cardiovascular disease (e.g. advanced heart failure, unstable angina, recent myocardial infarction, arrhythmias, uncontrolled hypertension or hypotension, aortic stenosis, thromboembolic events).
* Respiratory disorders (e.g. chronic respiratory failure or a moderate/severe BODEx index).
* Endocrine/metabolic diseases (e.g. uncontrolled diabetes).
* Neurological or psychiatric disorders (e.g. dementia).
* Prior use of ergogenic nutritional supplements.
* Any other condition deemed incompatible with moderate physical activity by the clinical team.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identified as women
Enrollment: 20 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Handgrip strength | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Handgrip strength (kg) was assessed with a digital handheld dynamometer (JAMAR®, 0-90 kg; Performance Health, Warrenville, IL, USA), by standardised procedures.
Cardiorespiratory | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Cardiorespiratory fitness was evaluated using the six-minute walk test (6MWT) on a standardised indoor 400-metre track.
Gait speed | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Gait speed was measured over four metres using photoelectric timing gates. Participants began walking five metres before the start line to ensure a consistent pace throughout the timed section.
Lower limb strength | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Lower limb strength was assessed using the Five Times Sit-to-Stand Test (5xSTS), which involved recording the time taken to rise from a 45 cm highchair five times as quickly as possible without using the arms for support.
Balance | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Balance was assessed via static balance testing in three different stances, held for 10 seconds each: side-by-side, semi-tandem and tandem
Frailty and global physical function | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Frailty and global physical function were evaluated using the Short Physical Performance Battery (SPPB), which incorporates tests of gait speed, balance, and the ability to rise from a chair. Based on the total score obtained in all tests (range from 0 to 10), participants are identified as having severe limitations (0-4), moderate limitations (4-6), mild limitations (7-9) and minimal limitations (10-12).
High-density lipoprotein (HDL) | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  High-density lipoprotein (HDL) was evaluated to explore potential cardiovascular implications.
  Venous blood samples were collected under standardised conditions between 08:00 and 08:30 a.m., following a minimum of 12 hours' fasting and at least eight hours' rest overnight. All extractions were performed by a certified nurse at an accredited clinical laboratory (Det Norske Veritas, certification no. 18031, Spain). A total of 10 ml of serum was drawn into clot-activator tubes, centrifuged and stored at -20 °C until analysis. Meanwhile, 3-5 mL of plasma was collected in EDTA® tubes and refrigerated at 4 °C for subsequent processing. All analytical procedures were conducted using standardised and validated platforms. Haematological assessments were performed using the Coulter Counter MAX-M® system, while biochemical and hormonal analyses were conducted using the Architect 2000® analyser (Abbott Diagnostics).
Creatine kinase | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Creatine kinase was measured as an indicator of muscle damage.
  Venous blood samples were collected under standardised conditions between 08:00 and 08:30 a.m., following a minimum of 12 hours' fasting and at least eight hours' rest overnight. All extractions were performed by a certified nurse at an accredited clinical laboratory (Det Norske Veritas, certification no. 18031, Spain).
  A total of 10 ml of serum was drawn into clot-activator tubes, centrifuged and stored at -20 °C until analysis. Meanwhile, 3-5 mL of plasma was collected in EDTA® tubes and refrigerated at 4 °C for subsequent processing.
  All analytical procedures were conducted using standardised and validated platforms. Haematological assessments were performed using the Coulter Counter MAX-M® system, while biochemical and hormonal analyses were conducted using the Architect 2000® analyser (Abbott Diagnostics).
Liver enzyme activity | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Liver enzyme activity was assessed via serum levels of aspartate aminotransferase (AST/GOT) and alanine aminotransferase (ALT/GPT).
  Venous blood samples were collected under standardised conditions between 08:00 and 08:30 a.m., following a minimum of 12 hours' fasting and at least eight hours' rest overnight. All extractions were performed by a certified nurse at an accredited clinical laboratory (Det Norske Veritas, certification no. 18031, Spain).
  A total of 10 ml of serum was drawn into clot-activator tubes, centrifuged and stored at -20 °C until analysis. Meanwhile, 3-5 mL of plasma was collected in EDTA® tubes and refrigerated at 4 °C for subsequent processing.
  All analytical procedures were conducted using standardised and validated platforms. Haematological assessments were performed using the Coulter Counter MAX-M® system, while biochemical and hormonal analyses were conducted using the Architect 2000® analyser (Abbott Diagnostics).
Low-density lipoprotein (LDL) | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Low-density lipoprotein (HDL) was evaluated to explore potential cardiovascular implications.
  Venous blood samples were collected under standardised conditions between 08:00 and 08:30 a.m., following a minimum of 12 hours' fasting and at least eight hours' rest overnight. All extractions were performed by a certified nurse at an accredited clinical laboratory (Det Norske Veritas, certification no. 18031, Spain). A total of 10 ml of serum was drawn into clot-activator tubes, centrifuged and stored at -20 °C until analysis. Meanwhile, 3-5 mL of plasma was collected in EDTA® tubes and refrigerated at 4 °C for subsequent processing. All analytical procedures were conducted using standardised and validated platforms. Haematological assessments were performed using the Coulter Counter MAX-M® system, while biochemical and hormonal analyses were conducted using the Architect 2000® analyser (Abbott Diagnostics).
Glucose | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Glucose provided insight into metabolic regulation. Venous blood samples were collected under standardised conditions between 08:00 and 08:30 a.m., following a minimum of 12 hours' fasting and at least eight hours' rest overnight. All extractions were performed by a certified nurse at an accredited clinical laboratory (Det Norske Veritas, certification no. 18031, Spain). A total of 10 ml of serum was drawn into clot-activator tubes, centrifuged and stored at -20 °C until analysis. Meanwhile, 3-5 mL of plasma was collected in EDTA® tubes and refrigerated at 4 °C for subsequent processing. All analytical procedures were conducted using standardised and validated platforms. Haematological assessments were performed using the Coulter Counter MAX-M® system, while biochemical and hormonal analyses were conducted using the Architect 2000® analyser (Abbott Diagnostics).
Testosterone | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Testosterone was used to evaluate the hormonal status and potential anabolic-catabolic shifts.
  Venous blood samples were collected under standardised conditions between 08:00 and 08:30 a.m., following a minimum of 12 hours' fasting and at least eight hours' rest overnight. All extractions were performed by a certified nurse at an accredited clinical laboratory (Det Norske Veritas, certification no. 18031, Spain). A total of 10 ml of serum was drawn into clot-activator tubes, centrifuged and stored at -20 °C until analysis. Meanwhile, 3-5 mL of plasma was collected in EDTA® tubes and refrigerated at 4 °C for subsequent processing. All analytical procedures were conducted using standardised and validated platforms. Haematological assessments were performed using the Coulter Counter MAX-M® system, while biochemical and hormonal analyses were conducted using the Architect 2000® analyser (Abbott Diagnostics).

SECONDARY OUTCOMES:
Quality of life questionnaire | At baseline, immediately before the start of the supplementation protocol, and at the end of the six-week intervention period, within 24 hours of the final exercise session
  Quality of life was measured using the World Health Organization Quality of Life Questionnaire - Brief Version (WHOQOL-BREF). The scale ranges from 0 to 100. Higher scores indicate a higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- City Council of Soria, Soria, Spain

IPD SHARING:
Plan to Share IPD: No